CLINICAL TRIAL: NCT06432855
Title: Genetic Determinants of the Antiviral Immune Response in Oceanian Populations
Acronym: GEDIPOP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-035; 2023-A02206-39 (Other: ID RCB)
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-05

CONDITIONS: Virus
Keywords: dengue; immunity; genetics; Ocenian populations; New Caledonia
MeSH Terms: conditions — Virus Diseases; Dengue | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-febrile adults of Melanesian and European origin (Other): Saliva samples and 20 mL blood samples from individuals of Melanesian and European origin from NC
  Interventions: Other: Blood collection; Other: saliva collection

INTERVENTIONS:
Other: Blood collection — 20 ml-blood sample
Other: saliva collection — saliva sample

SUMMARY:
Oceania's populations, including Melanesians, are paying a heavy price for dengue fever, which has been circulating actively in the region since the Second World War. In New Caledonia (NC), the incidence of dengue fever is higher among municipalities predominantly populated by Melanesians, suggesting that Melanesians may have an increased susceptibility to symptomatic dengue fever. Differences in antiviral immune responses between populations of different geographical origins are partly the result of population-specific immune regulatory variants. In turn, viruses have imposed considerable selective pressure on human populations. Although crucial to understanding their susceptibility to viral infections, the genetic determinants of the antiviral immune response of Oceanians remain to be characterized.

In this context, the hypothesis is that the genetic origin of Oceanians, and Melanesians in particular, has shaped their antiviral immune response and contributes to their greater susceptibility to certain viral infections. The aim is to characterize the immune response to pathogens affecting the New Caledonian population, and in particular to dengue virus, of Melanesian and European populations, and to identify its genetic determinants. It will be explored whether saliva can be used as a non-invasive sample to study the seroprevalence of dengue in Oceanian populations.

DETAILED DESCRIPTION:
Cross-sectional observational study with prospective sample and data collection Individuals will be identified from among eligible participants in the STEP-BSA21 and COVCAL studies.

Information and consent Questionnaire, saliva collection on Oragene tube, buccal swabbing and 20 mL blood collection on CPT tube

DNA extraction and low-coverage sequencing of participants' complete genomes And Isolation and in vitro stimulation of peripheral blood mononuclear cells (PBMCs) with dengue virus

* single-cell RNA sequencing (scRNAseq)
* multiplex quantification of cytokines and chemokines
* bioinformatics analysis to identify genetic markers associated with a differential transcriptomic and secretory response to dengue virus stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Non-febrile
* Self-declared member of the Melanesian or European community
* Having given consent to participate in the study

Exclusion Criteria:

* People who have taken part in a clinical study in the last 6 months in which they were exposed to a health product as part of the investigation (pharmaceutical product or device or placebo).
* People taking part in an ongoing clinical study
* People declaring themselves to belong to two communities (e.g. people of mixed European and Melanesian descent)
* Pregnant and breast-feeding women (in whom the immune response could be modified)
* People with a long-term medical condition (as defined by the French social security system) that could have an effect on the immune response, excluding dengue risk factors prevalent in New Caledonia such as diabetes, overweight/obesity and hypertension.
* Individuals with an acute infection (viral, bacterial or fungal) within 3 months of inclusion.
* Chronic administration (for more than 14 days) of immunosuppressants or treatments affecting the immune system in the 6 months prior to inclusion. For corticosteroids, this corresponds to a dose equivalent to 20 mg/day of prednisone or equivalent for more than two weeks (inhaled or topical steroids are permitted).
* Administration of a vaccine within 3 months prior to inclusion.
* Administration of blood products or immunoglobulins within 3 months of inclusion.
* People with known allergies to antibiotics, which could have an impact on the in vitro culture of PBMCs in the presence of antibiotics
* Persons not intellectually capable of answering the questionnaire
* Persons under guardianship, curatorship or any other legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Identify the genetic determinants of the innate immune response to pathogens affecting the New Caledonian population, and in particular to the dengue virus in individuals of Melanesian and European origin. | 3 years
  Identification by genomic techniques of expression Quantitative Trait Loci (eQTL) specifically associated with the innate immune response of Peripheral Blood Mononuclear Cells (PBMCs) collected from individuals of Melanesian and European origin and stimulated in vitro by DENV.

SECONDARY OUTCOMES:
To describe the genetic diversity of Melanesian and European populations in NC in relation to the determinants of susceptibility to health problems affecting NC populations. | 3 years
  Low-coverage DNA sequencing of the complete genome of individuals of Melanesian and European origin.
Characterizing the transcriptomic response to DENV in individuals of Melanesian and European origin. | 3 years
  Quantification by single cell RNAseq techniques of differentially expressed transcripts in response to in vitro dengue virus stimulation by Peripheral Blood Mononuclear Cells (PBMCs) collected from individuals of Melanesian and European origin.
Characterize the cytokine and chemokine response to DENV in individuals of Melanesian and European origin. | 3 years
  Quantification by multiplex techniques of the concentration of cytokines and chemokines differentially secreted in response to in vitro stimulation by dengue virus by Peripheral Blood Mononuclear Cells (PBMCs) collected from individuals of Melanesian and European origin.
Study the effect of environmental factors (smoking/non-smoking status, history of Cytomegalovirus or dengue virus infection, presence of diabetes, etc.) on the immune response to dengue virus. | 3 years
  Multivariate analyses of the association of environmental factors collected during the inclusion visit (questionnaire and measurements) or during analyses conducted as part of the present research with the immune response targeting the dengue virus.
Study the oral microbiome of individuals of Melanesian and European origin and analyze its association with the immune response to pathogens. | 3 years
  Next-generation sequencing and analysis of the oral microbiome on a saliva sample
Determine whether history of dengue virus infection can be demonstrated by testing saliva for antibodies using the Luminex technique. | 3 years
  Luminex quantification of dengue virus antibodies in serum and saliva from Melanesian and European individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Jouan, MD, Principal Investigator — Institut Pasteur de Nouvelle-Calédonie
Locations (1):
- Institut Pasteur de Nouvelle-Calédonie, Noumea, New Caledonia